CLINICAL TRIAL: NCT07292168
Title: A Phase 1b/2 Study Evaluating the Safety and Preliminary Efficacy of OM-RCA-01, an Anti-FGFR1 Monoclonal Antibody, in Patients With Metastatic Cancers Expressing FGFR1.
Brief Title: A Phase 1b/2 Study of the Safety and Efficacy of the Monoclonal Antibody OM-RCA-01 in Patients With Metastatic Tumors Expressing Fibroblast Growth Factor Receptor 1
Acronym: TAGNOT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMRCA01-TAGNOT
Record Dates: First submitted 2025-11-20; First posted 2025-12-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma Metastatic; Prostate Cancer Metastatic; Non-small Cell Lung Cancer Metastatic; Breast Cancer Metastatic; Head & Neck Cancer
Keywords: metastatic cancer; resistance; monoclonal antibody; fibroblast growth factor receptor 1; OM-RCA-01; kidney cancer; prostate cancer; head & neck cancer; lung cancer; breast cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis; Acrocephalosyndactylia; Kidney Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): OM-RCA-01
  Interventions: Biological: humanized monoclonal anti-FGFR1 antibody OM-RCA-01

INTERVENTIONS:
Biological: humanized monoclonal anti-FGFR1 antibody OM-RCA-01 — OM-RCA-01, solution for infusion, 25 mg/mL; 50 mg (dose level 1) or 100 mg (dose level 2), intravenously, every 14 days

SUMMARY:
One of the most relevant targets in the field of novel targeted anticancer therapy is the family of receptors to fibroblast growth factor receptors (FGFRs). FGFR1 is the main representative of the FGFR family.

The goal of this clinical trial is to learn if monoclonal anti-FGFR1 antibody (OM-RCA-01) works to treat metastatic cancers expressing FGFR1. It will also learn about the safety of drug OM-RCA-01. The main questions it aims to answer are:

1. What medical problems do participants have when receiving drug OM-RCA-01?
2. What dose of the drug should patients receive in the next studies?
3. Does tumor growth slow down in patients receiving OM-RCA-01?

All patients in this study will receive the antibody treatment. The drug will be given through a vein (by IV infusion) every two weeks, for as long as the disease remains under control and the treatment is well tolerated.

DETAILED DESCRIPTION:
FGFR1 is expressed on cells of various tumors, enabling their development. Currently, there are no reported monoclonal antibodies that block FGFR1, and only one chemically synthesized non-selective pan-FGFR inhibitor has been approved in the treatment of FGFR1-positive relapsed or refractory myeloid/lymphoid neoplasms.

OM-RCA-01 is an original innovative targeting drug focused on blocking FGFR1. OM-RCA-01 binds to the extracellular part of FGFR1. The main mechanism of action is blocking the activation processes of FGFR1. In studies, OM-RCA-01 was found to be a high-affinity and specific to FGFR1 antibody, inhibiting the phosphorylation of the receptor and the subsequent intracellular cascade. The amount of human protein in the structure of the humanized antibody is 92.9%.

The present clinical trial is a Phase 1b/2, multicenter, open-label, non-randomized, cohort study designed to evaluate the safety and preliminary efficacy of the monoclonal antibody OM-RCA-01 in patients with metastatic solid tumors expressing FGFR1.

This study adopts a basket trial design, enrolling patients based on the shared molecular characteristic of FGFR1 expression regardless of tumor histology. This approach enables the assessment of the anti-FGFR1 antibody's activity across multiple tumor types simultaneously.

Patients with FGFR1 expression meeting inclusion criteria (see the relevant section) will be enrolled into one of five tumor-specific cohorts:

* Renal cell carcinoma (RCC);
* Non-small cell lung cancer (NSCLC);
* Head and neck cancer (HNC);
* Breast cancer (BC);
* Prostate cancer (PCa) A total of 58 patients will be included. The study drug is administered intravenously, every 14 days till disease progression (RECIST 1.1) or unexaptable toxicity (CTCAE v.5.0).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form confirming voluntary participation in the study.
2. Age ≥ 18 years at the time of consent.
3. Body weight ≥ 50 kg.
4. Histologically confirmed metastatic solid tumors:

   1. clear-cell renal cell carcinoma;
   2. non-small cell lung cancer (adenocarcinoma or squamous cell cancer without EGFR and ALK mutations);
   3. prostate cancer (castration-resistant adenocarcinoma);
   4. breast cancer (adenocarcinoma with specified status for estrogen receptors, progesterone receptors, HER2);
   5. head and neck tumors (squamous carcinoma, salivary gland cancer).
5. Immunohistochemical expression of FGFR1 of 2+ or higher.
6. Documented disease progression after at least two lines of standard therapy, or lack of available or feasible alternative standard treatment options for any reason.
7. Presence of at least one measurable lesion according to RECIST 1.1 criteria.
8. Availability of formalin-fixed and paraffin-embedded tumor tissue samples for biomarker analysis.
9. ECOG performance status 0 or 1.
10. Adequate organ function, confirmed by laboratory test results obtained within 7 days prior to Cycle 1 Day 1, meeting the following parameters:

    * Hemoglobin level ≥ 90 g/L
    * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
    * Platelet count ≥ 100 × 10⁹/L
    * Serum creatinine level ≤ 1.5 × upper limit of normal (ULN)
    * Glomerular Filtration Rate (GFR) ≥ 30 mL/min
    * AST and ALT ≤ 3 × ULN (≤ 5 × ULN in patients with liver metastases)
    * Serum phosphorus within normal limits (≥ lower limit of normal and ≤ upper limit of normal)
    * Serum calcium ≥ lower limit of normal
    * Serum potassium ≥ lower limit of normal (note: use of medications to increase potassium during screening is permitted)
11. Life expectancy of more than 12 weeks.
12. Absence of any psychological, familial, social or geographical circumstances that could potentially serve as an obstacle to the fulfillment of the study protocol and follow-up procedures according to the prescribed schedule and the ability of the study participant to follow the requirements of the protocol; these circumstances should be discussed with the patient before inclusion in the study.
13. Women capable of childbearing must be using an effective method of contraception.

Exclusion Criteria:

1. Participation in another clinical trial or concomitant treatment with any investigational drug, or administration of any investigational anticancer therapy within 28 days prior to inclusion in this study.
2. Presence of central nervous system (CNS) metastases and/or medullary carcinomatosis at the time of inclusion.

   Exception: Patients with CNS metastases who have received therapy may participate if they have been clinically stable for at least 1 month prior to enrollment, defined by:
   * No evidence of new or progressive CNS metastases
   * No ongoing steroid therapy
   * Stable mental status sufficient to provide informed consent
3. History of or current evidence of any condition, therapy, or laboratory abnormality that could:

   * Limit interpretation of study results,
   * Prevent completion of the study protocol, or
   * Pose a risk to patient safety or well-being. This includes any serious or unstable general medical, psychiatric, or other conditions potentially jeopardizing safety, informed consent, or compliance.
4. Any second malignancy within the previous 5 years, except for adequately treated cervical carcinoma in situ, squamous cell carcinoma of the skin, or basal cell carcinoma of the skin with limited growth, provided these are well controlled.
5. Known regular use of illicit substances or recreational drugs, or a history of drug abuse or alcoholism within the past year.
6. Plans to conceive during the study period, current pregnancy, or lactation.
7. Known HIV-positive status.
8. Known active hepatitis B or C infection.
9. Evidence of active bleeding or hemorrhagic diathesis.
10. Radiation therapy within 14 days prior to inclusion.
11. Receipt of any anti-tumor treatments including:

    * Surgery or tumor embolization within 14 days prior to the first OM-RCA-01 dose, or
    * Chemotherapy, immunotherapy, biological therapy, investigational therapy, or endocrine therapy (except ongoing androgen deprivation therapy for prostate cancer) within 14 days or within two half-lives of the drug (whichever is longer) prior to the first OM-RCA-01 dose.
12. Prior treatment with any FGFR-inhibiting or FGFR-blocking agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint in the phase 1b study | 6 months
  Recommended Phase 2 Dose (RP2D)
Primary endpoint in the phase 2 study | 12 months
  Objective response rate according to RECIST 1.1 criteria as assessed by the investigator

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events (AEs) as Assessed by CTCAE v5.0 | 12 months
Number of Participants with serious AEs | 12 months
Median progression-free survival | 12 months
12-month progression-free survival rate | 12 months
Median overall survival | 12 months
12-month overall survival rate | 12 months
Median duration of response | 12 months
Quality of life, assessed using the EORTC QLQ-C30 questionnaire | 8 weeks
  in patients before and after 8 weeks of therapy (0-100)
Concentration of anti-drug antibodies | 12 months
  Assessment of immunogenicity
Pharmacokinetics profile: Cmax | 1 month
  the highest concentration of OM-RCA-01 in the blood
Pharmacokinetics profile: Tmax | 1 month
  The time it takes for a antibody to reach the maximum concentration
Pharmacokinetics profile: AUC0-t | 1 month
  the area under the plasma concentration-time curve from time zero to time t
Pharmacokinetics profile: CL | 1 month
  clearance
Pharmacokinetics profile: T1/2 | 1 month
  the time required for plasma concentration of a OM-RCA-01 to decrease by 50%
Pharmacokinetics profile: Vss | 1 month
  Steady-state volume of distribution
Pharmacokinetics profile: Kel | 1 month
  the elimination rate constant

OTHER OUTCOMES:
Analysis of objective response rate, progression-free survival and overall survival based on FGFR1 expression level | 12 months
  FGFR1 immunohistochemical expression (IHC) 3+ versus IHC 2+ in tumors;
Assessment of Biomarkers: cfDNA | 12 months
  cfDNA level in plasma
Assessment of Biomarkers: sFlt-1 | 12 months
  sFlt-1 in plasma

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - Republican Dispensary of Tatarstan, Kazan'
  - A.I. Kryzhanovsky Krasnoyarsk Regional Cancer Center, Krasnoyarsk
  - Hadassah Medical, Moscow
  - I.P. Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Republican Clinical Oncology Dispensary, Ufa

IPD SHARING:
Plan to Share IPD: Undecided